CLINICAL TRIAL: NCT02031159
Title: Correlation, Accuracy, Precision and Practicability of Zero Heat Flux Method in Comparison With Sublingual and Nasopharyngeal Temperature Measurement
Brief Title: Correlation, Accuracy, Precision and Practicability of Zero Heat Flux Temperature Monitoring
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, PD Dr. Jan Hoecker, PD Dr. Jan Höcker, University Hospital Schleswig-Holstein
Other Study IDs: THER-ZeroHeatFlux
Record Dates: First submitted 2014-01-01; First posted 2014-01-09 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Hypothermia
Keywords: perioperative hypothermia; zero heat flux; non-invasive measurement of body core temperature
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hypothermia is common in patients undergoing general anesthesia. There have been several negative outcomes reported. Zero heat flux is a non-invasive method for measurement of body core temperature. The aim of this study is to see if this method is comparable in terms of correlation, accuracy, precision and practicability to commonly used sublingual and nasopharyngeal temperature monitoring.

DETAILED DESCRIPTION:
Hypothermia is common in patients undergoing general anesthesia. There have been several negative outcomes reported such as bleeding, infection rate, cardiac complications, prolonged wound healing and patient discomfort. Zero heat flux is a non-invasive method for measurement of body core temperature. The aim of this study is to see if this method is comparable in terms of correlation, accuracy, precision and practicability to commonly used sublingual and nasopharyngeal temperature monitoring. Measurements are performed with the SpotOn® sensor by Arizant Healthcare, Inc..

ELIGIBILITY:
Inclusion Criteria:

* elective surgery in gynecology or trauma surgery
* planned surgery time > 60 min
* patients older than 16 years

Exclusion Criteria:

* emergency surgery
* need for post-surgery ventilation
* patient's denial to take part in the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 16 years undergoing elective surgery in either gynecology or trauma surgery with a planned surgery time > 60 min.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
body core temperature (°C) | body core temperature taken at 15 min after induction of anesthesia

SECONDARY OUTCOMES:
body core temperature (°C) | body core temperature taken at 45 min after induction of anesthesia

OTHER OUTCOMES:
body core temperature (°C) | body core temperature taken at 75 min after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hoecker, MD, Study Director — Klinik fur Anästhesiologie und Operative Intensivmedizin
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Anästhesiologie und Operative Intensivmedizin, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Teunissen LP, Klewer J, de Haan A, de Koning JJ, Daanen HA. Non-invasive continuous core temperature measurement by zero heat flux. Physiol Meas. 2011 May;32(5):559-70. doi: 10.1088/0967-3334/32/5/005. Epub 2011 Mar 28. PMID 21444968
- [Derived] Iden T, Horn EP, Bein B, Bohm R, Beese J, Hocker J. Intraoperative temperature monitoring with zero heat flux technology (3M SpotOn sensor) in comparison with sublingual and nasopharyngeal temperature: An observational study. Eur J Anaesthesiol. 2015 Jun;32(6):387-91. doi: 10.1097/EJA.0000000000000232. PMID 25693138